CLINICAL TRIAL: NCT01579617
Title: e-SiHLE: An Internet Pregnancy Prevention for Older Teenage Girls
Acronym: eSiHLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patricia Kissinger, Professor, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 261904-1; TP2AH000013 (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2012-03-06; First posted 2012-04-18 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Pregnancy; Sexually Transmitted Infections
Keywords: pregnancy; STI; STD
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BUtiful (Experimental): Intervention arm, 'BUtiful. Be yoU! Talented, Informed, Fearless, Uncompromised, Loved', has 8 website sessions focused on pregnancy and STI prevention
  Interventions: Behavioral: BUtiful.
- DIVAS (Other): Attention control arm, 'DIVAS. Diversity, Individuality, Vitality, Activity and Strong', has 8 website sessions focused on general health and nutrition
  Interventions: Behavioral: DIVAS.

INTERVENTIONS:
Behavioral: BUtiful. — 8 website sessions include themes that teach: gender empowerment, assertive communication skills, goal setting, pregnancy and STI/HIV risk, safer sex behaviors, proper condom use, positive attitudes and norms towards consistent condom use, contraception, partner involvement in safer sex, and responsibility for their own health.
  Other Names: BUtiful
  Arms: BUtiful
Behavioral: DIVAS. — Attention control arm: 8 website sessions that include topics on: healthy eating, choosing nutritional snacks, sugar and salt intake, physical activity, stress management, foods for beauty.
  Other Names: DIVAS
  Arms: DIVAS

SUMMARY:
The purpose of this study is to evaluate the efficacy of an online pregnancy prevention intervention that was adapted from the evidence based small group intervention SiHLE.

DETAILED DESCRIPTION:
The investigators will test the hypothesis that by the end of the study, women who receive the e-SIHLE intervention will have a 35% increase in reliable contraception use compared to attention control website, DIVAS, which is a health and nutrition education program.

Both arms of the study were designed for African-American women who are 18-19 years old.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or 19 at enrollment
* Female
* Not currently pregnant or intending to become pregnant in the next 12 months
* Live in Orleans or Jefferson Parish in Louisiana
* English is your primary language
* Access to a computer and internet connection
* Does not have sex with women exclusively

Exclusion Criteria:

* Age younger than 18 or older than 19
* Male
* Currently pregnant or intend to become pregnant in the next 12 months
* Live outside of Orleans or Jefferson Parish
* Hearing impairments that prevent listening to videos

Ages: 18 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 637 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in the use of reliable contraceptives | Change from baseline measured at 3 and 7 and 13 months post baseline
  Women who receive the BUtiful intervention will have a 35% increase in the use of reliable contraceptives compared to the DIVAS intervention. Reliable contraceptive use is defined as the consistent use of a condom with all sex partners, a hormonal birth control method, or an intrauterine device.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kissinger, BSN MPH PhD, Principal Investigator — Tulane University Health Sciences Center, School of Public Health and Tropical Medicine
Locations (6):
- United States (6):
  - Community Intercept, New Orleans, Louisiana
  - Tulane Drop In Clinic at Covenant House, New Orleans, Louisiana
  - Delgado Community College, New Orleans, Louisiana
  - Dillard University, New Orleans, Louisiana
  - Xavier University, New Orleans, Louisiana
  - Southern University of New Orleans, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh S, Darroch JE. Adolescent pregnancy and childbearing: levels and trends in developed countries. Fam Plann Perspect. 2000 Jan-Feb;32(1):14-23. PMID 10710702
- [Background] Kost, K., Henshaw, S., & Carlin, L. , U.S. Teenage Pregnancies, Births and Abortions: National and State Trends and Trends by Race and Ethnicity. . 2010, Guttmacher: New York.
- [Background] Guttmacher Institute, Facts on American Teens' Sexual and Reproductive Health. 2010, Guttmacher Institute New York.
- [Background] Guttmacher Institute, U.S. Teenage Pregnancy Statistics: National and State Trends and Trends by Race and Ethnicity. . 2006, Guttmacher Institute: New York.
- [Background] Prevention, C.f.D.C.a., Youth Risk Behavior Surveillance Survey. 2007, Centers for Disease Control and Prevention
- [Background] Hamilton, B.E., Martin, J. A., & Ventura, S. J., National Vital Statistics Reports. 2007, Centers for Disease Control and Prevention.
- [Background] Mosher WD, Martinez GM, Chandra A, Abma JC, Willson SJ. Use of contraception and use of family planning services in the United States: 1982-2002. Adv Data. 2004 Dec 10;(350):1-36. PMID 15633582
- [Background] Foundation, T.A.E.C., Kids Count 2008 data book 2008, The Annie E. Casey Foundation Baltimore.
- [Background] Frost JJ, Darroch JE. Factors associated with contraceptive choice and inconsistent method use, United States, 2004. Perspect Sex Reprod Health. 2008 Jun;40(2):94-104. doi: 10.1363/4009408. PMID 18577142
- [Background] Finer LB, Henshaw SK. Disparities in rates of unintended pregnancy in the United States, 1994 and 2001. Perspect Sex Reprod Health. 2006 Jun;38(2):90-6. doi: 10.1363/psrh.38.090.06. PMID 16772190
- [Background] Zill, N., & O'Donnell, K., Child poverty rates by maternal risk factors: An update. 2004, WESTAT.
- [Background] Martin JA, Hamilton BE, Sutton PD, Ventura SJ, Menacker F, Kirmeyer S, Munson ML; Centers for Disease Control and Prevention National Center for Health Statistics National Vital Statistics System. Births: final data for 2005. Natl Vital Stat Rep. 2007 Dec 5;56(6):1-103. PMID 18277471
- [Background] Hoffman, S.D., By the numbers: The public costs of adolescent childbearing. 2006, The National Campaign to Prevent Teen Pregnancy.: Washington, DC.
- [Background] The National Campaign to Prevent Teen Pregnancy, Why it matters: Linking teen pregnancy prevention to other critical social issues. 2010: Washington, DC.
- [Background] Kissinger P, Clark R, Rice J, Kutzen H, Morse A, Brandon W. Evaluation of a program to remove barriers to public health care for women with HIV infection. South Med J. 1995 Nov;88(11):1121-5. doi: 10.1097/00007611-199511000-00007. PMID 7481982
- [Background] Bedimo AL, Bessinger R, Kissinger P. Reproductive choices among HIV-positive women. Soc Sci Med. 1998 Jan;46(2):171-9. doi: 10.1016/s0277-9536(97)00157-3. PMID 9447641
- [Background] Fuller C, Clark RA, Kissinger P, Abdalian SE. Clinical manifestations of infection with human immunodeficiency virus among adolescents in Louisiana. J Adolesc Health. 1996 Jun;18(6):422-8. doi: 10.1016/1054-139X(95)00235-K. PMID 8803734
- [Background] Bessinger R, Clark R, Kissinger P, Rice J, Coughlin S. Pregnancy is not associated with the progression of HIV disease in women attending an HIV outpatient program. Am J Epidemiol. 1998 Mar 1;147(5):434-40. doi: 10.1093/oxfordjournals.aje.a009468. PMID 9525529
- [Background] Kissinger P, Fuller C, Clark RA, Abdalian SE. Psychosocial characteristics of HIV-infected adolescents in New Orleans. J Adolesc Health. 1997 Apr;20(4):258. doi: 10.1016/S1054-139X(97)00029-3. No abstract available. PMID 9098727
- [Background] Kissinger P, Mohammed H, Richardson-Alston G, Leichliter JS, Taylor SN, Martin DH, Farley TA. Patient-delivered partner treatment for male urethritis: a randomized, controlled trial. Clin Infect Dis. 2005 Sep 1;41(5):623-9. doi: 10.1086/432476. Epub 2005 Jul 19. PMID 16080084
- [Background] Kissinger P, Schmidt N, Mohammed H, Leichliter JS, Gift TL, Meadors B, Sanders C, Farley TA. Patient-delivered partner treatment for Trichomonas vaginalis infection: a randomized controlled trial. Sex Transm Dis. 2006 Jul;33(7):445-50. doi: 10.1097/01.olq.0000204511.84485.4c. PMID 16531939
- [Background] Schillinger JA, Kissinger P, Calvet H, Whittington WL, Ransom RL, Sternberg MR, Berman SM, Kent CK, Martin DH, Oh MK, Handsfield HH, Bolan G, Markowitz LE, Fortenberry JD. Patient-delivered partner treatment with azithromycin to prevent repeated Chlamydia trachomatis infection among women: a randomized, controlled trial. Sex Transm Dis. 2003 Jan;30(1):49-56. doi: 10.1097/00007435-200301000-00011. PMID 12514443
- [Background] Kissinger P, Brown R, Reed K, Salifou J, Drake A, Farley TA, Martin DH. Effectiveness of patient delivered partner medication for preventing recurrent Chlamydia trachomatis. Sex Transm Infect. 1998 Oct;74(5):331-3. doi: 10.1136/sti.74.5.331. PMID 10195027
- [Background] Kissinger, P., et al. Recurrent Trichomonas vaginalis among HIV positive and negative women. in 16th ISSTDR. 2005. Amsterdam, Netherlands.
- [Background] Kissinger P, Amedee A, Clark RA, Dumestre J, Theall KP, Myers L, Hagensee ME, Farley TA, Martin DH. Trichomonas vaginalis treatment reduces vaginal HIV-1 shedding. Sex Transm Dis. 2009 Jan;36(1):11-6. doi: 10.1097/OLQ.0b013e318186decf. PMID 19008776
- [Background] Kissinger P, Secor WE, Leichliter JS, Clark RA, Schmidt N, Curtin E, Martin DH. Early repeated infections with Trichomonas vaginalis among HIV-positive and HIV-negative women. Clin Infect Dis. 2008 Apr 1;46(7):994-9. doi: 10.1086/529149. PMID 18444815
- [Background] Chaturvedi AK, Dumestre J, Gaffga AM, Mire KM, Clark RA, Braly PS, Dunlap K, Beckel TE, Hammons AF, Kissinger PJ, Hagensee ME. Prevalence of human papillomavirus genotypes in women from three clinical settings. J Med Virol. 2005 Jan;75(1):105-13. doi: 10.1002/jmv.20244. PMID 15543579
- [Background] Magnus M, Schillinger JA, Fortenberry JD, Berman SM, Kissinger P. Partner age not associated with recurrent Chlamydia trachomatis infection, condom use, or partner treatment and referral among adolescent women. J Adolesc Health. 2006 Sep;39(3):396-403. doi: 10.1016/j.jadohealth.2006.01.005. Epub 2006 Jul 10. PMID 16919802
- [Background] Kissinger P, Clark R, Dumestre J, Bessinger R. Incidence of three sexually transmitted diseases during a safer sex promotion program for HIV-infected women. J Gen Intern Med. 1996 Dec;11(12):750-2. doi: 10.1007/BF02598989. PMID 9016422
- [Background] Yoo S, Johnson CC, Rice J, Manuel P. A qualitative evaluation of the Students of Service (SOS) program for sexual abstinence in Louisiana. J Sch Health. 2004 Oct;74(8):329-34. doi: 10.1111/j.1746-1561.2004.tb06623.x. PMID 15554119
- [Background] Card JJ, Kuhn T, Solomon J, Benner TA, Wingood GM, DiClemente RJ. Translating an effective group-based HIV prevention program to a program delivered primarily by a computer: methods and outcomes. AIDS Educ Prev. 2011 Apr;23(2):159-74. doi: 10.1521/aeap.2011.23.2.159. PMID 21517664
- [Background] Latham TP, Sales JM, Boyce LS, Renfro TL, Wingood GM, DiClemente RJ, Rose E. Application of ADAPT-ITT: adapting an evidence-based HIV prevention intervention for incarcerated African American adolescent females. Health Promot Pract. 2010 May;11(3 Suppl):53S-60S. doi: 10.1177/1524839910361433. PMID 20488969
- [Background] Wingood GM, DiClemente RJ. The ADAPT-ITT model: a novel method of adapting evidence-based HIV Interventions. J Acquir Immune Defic Syndr. 2008 Mar 1;47 Suppl 1:S40-6. doi: 10.1097/QAI.0b013e3181605df1. PMID 18301133
- [Background] DiClemente RJ, Wingood GM, Harrington KF, Lang DL, Davies SL, Hook EW 3rd, Oh MK, Crosby RA, Hertzberg VS, Gordon AB, Hardin JW, Parker S, Robillard A. Efficacy of an HIV prevention intervention for African American adolescent girls: a randomized controlled trial. JAMA. 2004 Jul 14;292(2):171-9. doi: 10.1001/jama.292.2.171. PMID 15249566